CLINICAL TRIAL: NCT01799967
Title: Functional Assessment Following Minimally Invasive Surgery of the Gastro-Esophageal Junction
Brief Title: Minimally Invasive Surgery of the Gastro-esophageal Junction
Acronym: MISGEJ
Status: Active, not recruiting | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 2007173-01H
Record Dates: First submitted 2013-02-25; First posted 2013-02-27 (Estimated); Last update posted 2026-01-30 (Actual); Status verified 2024-12

CONDITIONS: Achalasia; Paraesophageal Hernia; GERD; Epiphrenic Diverticula; Zenker's Diverticulum
Keywords: gastro-esophageal junction; minimally invasive; Achalasia; Paraesophageal hernia; GERD; Epiphrenic diverticula; Zenker's diverticulum; All minimally invasive surgeries of the gastro-esophageal junction
MeSH Terms: conditions — Esophageal Achalasia; Hernia, Hiatal; Gastroesophageal Reflux; Zenker Diverticulum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will assess short and long term outcomes of individuals undergoing minimally invasive surgery of the gastro-esophageal junction (MISGEJ). Patients will respond to questionnaires on an annual basis evaluating quality of life and functionality following MISGEJ. Hospital charts will also be reviewed on an annual basis to assess patient health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All patients at the Ottawa Hospital undergoing minimally invasive surgery of the GEJ

Exclusion Criteria:

* Less than 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing minimally invasive surgery of the gastro-esophageal junction at the Ottawa Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2007-11; Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
MISGEJ symptoms (subjective) | 8 years
  MISGEJ symptom questionnaire evaluated on an annual basis
Achalasia Disease Severity (subjective) | 8 years
  Achalasia Disease Severity questionnaire evaluated on an annual basis.
Diagnostic imaging | 8 years
  Patient x-rays, upper GI tests, Endoscopy, and/or CT scans will be assessed on an annual basis to objectively measure functionality and health status.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew JE Seely, MD, PhD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- Ottawa Hospital Research Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided